CLINICAL TRIAL: NCT02314507
Title: Effects of Gua Sha and Hot Pack for Relieving Chronic Low Back Pain in Elderly: A Crossover Randomized Controlled Trial
Brief Title: Gua Sha for Chronic Low Back Pain in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John Yuen, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GS-001
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Back Pain
Keywords: Gua sha
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gua sha (Experimental): Paritcipants in this group will receive a single treatment of Gua sha conducted by a well-trained nurse or Chinese practitioner
  Interventions: Other: Gua sha
- Hot Pack Therapy (Active Comparator): Participants in this group will receive a single treatment of Hot Pack conducted by a well-trained nurse or Physiotherapist
  Interventions: Other: Hot pack

INTERVENTIONS:
Other: Gua sha — A smooth, rounded-edged Gua sha tool will be press-stroked into the flesh enough to contact the fascial layer start at the midline of the subject's back. A stroke line is typically 4 to 6 inches long. Press-stroking will be repeated in one direction until the petechiae raises on that stroke line, typically 8 to 12 strokes. Gua sha will then be continued at the next stroke line directly adjacent to the one before, until the area covered the lower one third of the back.
  Other Names: Skin scraping
  Arms: Gua sha
Other: Hot pack — A hydrocollator pack will be used and it will be stored at 42-43oC in the hydrocollator. 6 layers of towel will be used to cover the hydrocollator pack when applying to the back of the subjects.
  Arms: Hot Pack Therapy

SUMMARY:
The purpose of the study is to investigate whether Gua sha is an effective modality for relieving chronic low back pain specifically in the aged population by comparing the baseline measures of pain intensity, self-perceived disability, back range of motion, back local muscle stiffness, depression, sleeping quality, quality of life, biomarkers measurement, and analgesic intake on days 1 and 7 after a single session of Gua sha treatment. In addition, the investigators are going to compare between Gua sha and hot pack treatments for the above parameters.

DETAILED DESCRIPTION:
Subjects will be randomized to receive firstly either one of the treatment arms, and then crossed over to receive another arm after 30 days washing out period. It is expected that Gua sha is 1) effective in reducing the intensity of chronic low back pain in the elderly; 2) effective in helping one or more outcome measures in this study and 3) more effective on relieving the low back pain than hot pack in terms of the outcome measures in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or above
* Self-reported painful restriction of lumbar spine mobility for at least 3 months or self-reported low back pain on at least 5 days a week for at least 3 months
* Have pain intensity score 40 or above on a 100mm Visual Analog Scale (VAS) at baseline

Exclusion Criteria:

* Prior history of radiculopathy or spinal stenosis or spinal fusion or failed surgery syndrome
* Having radiating pain below the knee
* Received the following surgery at the region of treatment in the past 12 months laminectomy, laminotomy or discectomy
* Serious illness (e.g. malignancy)
* Having wounds or skin lesions at the region of treatment
* Having blood pressure at140/90 mmHg or above at baseline
* Having Body Mass Index (BMI) at 18.5 or lower at baseline (as calculated by the weight in kilograms divided by the square of the height in metres (kg/m2)
* Having active psychiatric disorders, significant mood disorder or dementia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Day 0 before treatment, Day 1 and day 7 after treatment
  Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Back range of motion | Day 0 before treatment, Day 1 and day 7 after treatment
  By using inclinometer
Biomarkers for inflammation and anti-inflammation | Day 0 before treatment, day 7 after treatment
  Saliva specimen is collected from each subject for measuring the levels of Tumor
Self-perceived disability | Day 0 before treatment, Day 1 and day 7 after treatment
  Roland-Morris Disability Questionnaire (RMDQ)
Depression level | Day 0 before treatment, Day 1 and day 7 after treatment
  Geriatric Depression Scale (GDS)
Sleeping quality | Day 0 before treatment, Day 1 and day 7 after treatment
  Pittsburgh Sleep Quality index (PSQI)
Quality of life | Day 0 before treatment, day 7 after treatment
  Short-Form (12) Questionnaire (SF-12)
Record for oral intake of NSAIDs and analgesic drugs | Day 0 before treatment, day 7 after treatment
  Record

CONTACTS AND LOCATIONS:
Overall Officials: John Yuen, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Kowloon, Hong Kong